CLINICAL TRIAL: NCT04797247
Title: Study to Evaluate the Long-Term Efficacy and Safety of LIB003 in Patients With Cardiovascular Disease on Stable Lipid-Lowering Therapy Requiring Additional LDL-C Reduction
Brief Title: Study of Efficacy and Safety of LIB003 in Patient With CVD on Statins Requiring Additional LDL-C Reduction
Acronym: LIBerate-CVD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LIB Therapeutics LLC (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIB003-005
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases; Hyper-LDL-cholesterolemia
Keywords: lerodalcibep; PCSK9 inhibitor
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: participants, study staff, investigator and sponsor blinded to treatment and lipid levels
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LIB003 (lerodalcibep) (Experimental): 300 mg subcutaneously monthly (Q4W)
  Interventions: Drug: lerodalcibep
- Placebo (Placebo Comparator): matching placebo subcutaneously monthly (Q4W)
  Interventions: Drug: lerodalcibep

INTERVENTIONS:
Drug: lerodalcibep — PCSK9 inhibitor
  Other Names: LIB003

SUMMARY:
This study is to assess LDL-C reductions at Week 52 with monthly (Q4W [≤31 days]) dosing of LIB003 (lerodalcibep) 300 mg administered subcutaneously (SC) compared to placebo in patients with very-high risk for CVD on a stable diet and oral LDL-C lowering drug therapy.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, Phase 3 study of 52 weeks duration.

Patients who fulfill the inclusion and exclusion criteria will be enrolled at up to 60 sites in the United States, Canada, Europe, South Africa, Asia, Australasia, and the Middle East. Patients will be randomized in a 2:1 ratio to LIB003 or placebo. The total study duration will be up to 63 weeks which includes up to a Screening Period and 52 weeks of study drug treatment. Following randomization patients will be dosed and seen in the clinic Q4W (≤31 days).

ELIGIBILITY:
Inclusion Criteria:

* Provision of written and signed informed consent prior to any study-specific procedure;
* Male or female ≥18 years of age at the first Screening Visit;
* Weight of ≥40 kg (88 lb) and body mass index (BMI) ≥17 and ≤42 kg/m2;
* At very high risk for CVD which includes history of CVD, (including cerebrovascular or peripheral arterial disease) or very high risk as defined in the 2019 ESC/EAS Guidelines
* At Screening or post Washout/Stabilization), ≥70 mg/dL and TG ≤400 mg/dL while on stable lipid-lowering oral drug therapy (i.e., maximally tolerated statin with or without ezetimibe); Patients unable to tolerate approved doses of a statin may take lower than approved doses and dose less frequently than daily as long as the dose and dosing frequency is consistent; Patients with documentation of inability to tolerate any statin at any dose, or history of rhabdomyolysis, may also participate;
* On a stable diet and lipid-lowering oral therapies (such as statins, ezetimibe, bile-acid sequestrants, OM-3 compounds, fenofibrate, bezafibrate, nicotinic acid, and bempedoic acid) or combinations thereof for at least 4 weeks
* Patients on a PCSK9 mAb at a dose of 75 mg, 140 mg, or 150 mg Q2W must undergo a washout period of ≥4 weeks after the last dose; for those on 300 mg or 420 mg Q4W (≤31 days) the washout period is ≥8 weeks following last dose; 8. Females of childbearing potential must be using a highly effective form of birth control if sexually active and have a negative urine pregnancy test at the last Screening Visit;

Exclusion Criteria:

* Use of prohibited oral lipid-lowering agents mipomersen or lomitapide within 6 months of screening, gemfibrozil within 6 weeks of screening, LDL or plasma apheresis within 2 months prior to randomization; received other investigational agent(s) such as PCSK9 or Lp(a) siRNA or locked nucleic acid-reducing agents within 12 months of the Screening Visit;
* Documented history of HoFH defined clinically or genetically
* History of any prior or active clinical condition or acute and/or unstable systemic disease compromising patient inclusion, at the discretion of the Investigator
* Females of childbearing potential who are sexually active, not using or unwilling to use a highly effective form of contraception, pregnant or breastfeeding, or who have a positive urine pregnancy test at the last Screening Visit;
* Moderate to severe renal dysfunction, defined as an eGFR <30 mL/min/1.73m2
* Active liver disease or hepatic dysfunction, history of liver transplant, and/or ALT or AST >2.5 × the ULN as determined by central laboratory analysis at screening
* Uncontrolled thyroid disease: hyperthyroidism or hypothyroidism 9. Uncontrolled Type 1 or Type 2 DM, defined as FBS ≥200 mg/dL or HbA1C ≥9%; 10. Uncontrolled serious cardiac arrhythmia, MI, unstable angina, PCI, CABG, placement of implantable cardioverter defibrillator or biventricular pacemaker, aortic valve surgery, or stroke within 3 months prior to the Screening Visit; 11. Planned cardiac surgery or revascularization; 12. New York Heart Association class III-IV heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
LDL-C change compared to placebo | 52 weeks
  Percent change in LS mean from baseline compared to placebo in LDL-C level
mean LDL-C change at week 50 and 52 | 52 weeks
  Percent change in LS mean from baseline compared to placebo in LDL-C level at Weeks 50 and 52

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by Medical Dictionary for Regulatory Activities as severe, moderate or mild after 52 weeks | 52 weeks
  Evaluation of Adverse Events based on MedRA based on ITT population
Free PCSK9 change | 52 weeks
  Percent change in LS mean from baseline compared to placebo in free PCSK9
Percentage of patients achieving 2019 ESC/EAS LDL-C goals | 52 weeks
  To assess the effects of LIB003 on the percentage of patients achieving an LDL-C <40 mg/dL, 55 mg/dL, <70 mg/dL, and 100 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Evan A Stein, MD PhD, Study Director — LIB Therapeutics
Locations (3):
- United States (3):
  - Sterling Research Group, Cincinnati, Ohio
  - The Lindner Research Center, Cincinnati, Ohio
  - Metabolic & Atherosclerosis Research Center (MARC), Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No